CLINICAL TRIAL: NCT06662396
Title: A Study to Evaluate the Effects of Coadministration of Diltiazem on the Plasma Pharmacokinetics of a Single Dose of MK-6552 in Healthy Participants
Brief Title: A Study of Diltiazem With a Single Dose of MK-6552 in Healthy Adult Participants (MK-6552-007)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6552-007; MK-6552-007 (Other: MSD)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-6552 + Diltiazem (Experimental): Participants receive a single dose of MK-6552 on Period 1 Day 1. Participants receive a Diltiazem every day (QD) for 6 days (Period 2 Days 1-6). On Period 2 Day 2 participants receive a single dose of MK-6552.
  Interventions: Drug: MK-6552; Drug: Diltiazem

INTERVENTIONS:
Drug: MK-6552 — Oral Gelatin Coated Capsule
Drug: Diltiazem — Oral Extended-Release Capsule

SUMMARY:
The main goal of this study is to learn what happens to MK-6552 in a person's body over time (a pharmacokinetic or PK study). Researchers want to know what happens to MK-6552 in healthy adults when a single dose of MK-6552 is given with multiple doses of diltiazem. The researchers believe that multiple doses of diltiazem will not affect the highest amount of MK-6552 in the blood.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Body Mass Index (BMI) between 18 and 32 kg/m^2, inclusive

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* History of cancer (malignancy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of MK-6552 | Pre-dose and at designated time points up to 24 hours post dose
  Blood samples will be collected to determine the Cmax of MK-6552 in plasma.

SECONDARY OUTCOMES:
Number of Participants Who Experience and Adverse Event (AEs) | Up to approximately 20 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 20 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) of MK-6552 | Pre-dose and at designated time points up to 96 hours post dose
  Blood samples will be collected to determine the AUC0-inf of MK-6552 in plasma.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24) of MK-6552 | Pre-dose and at designated time points up to 24 hours post dose
  Blood samples will be collected to determine the AUC0-24 of MK-6552 in plasma.
Time to Maximum Plasma Concentration (Tmax) of MK-6552 | Pre-dose and at designated time points up to 96 hours post dose
  Blood samples will be collected to determine the Tmax of MK-6552 in plasma.
Concentration of MK-6552 at 6 Hours Postdose (C6h) | Pre-dose and at designated time points up to 6 hours post dose
  Blood samples will be collected to determine the C6h of MK-6552 in plasma.
Concentration of MK-6552 at 8 Hours Postdose (C8h) | Pre-dose and at designated time points up to 8 hours post dose
  Blood samples will be collected to determine the C8h of MK-6552 in plasma.
Apparent Clearance (CL/F) of MK-6552 | Pre-dose and at designated time points up to 96 hours post dose
  Blood samples will be collected to determine the CL/F of MK-6552 in plasma.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-6552 | Pre-dose and at designated time points up to 96 hours post dose
  Blood samples will be collected to determine the Vz/F of MK-6552 in plasma.
Apparent Terminal Half-Life (t1/2) of MK-6552 | Pre-dose and at designated time points up to 96 hours post dose
  Blood samples will be collected to determine the t1/2 of MK-6552 in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- ICON (Site 0001), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com